CLINICAL TRIAL: NCT04137796
Title: Breastfeeding Behavior, Infant and Child Nutrition in Austria
Brief Title: Infant Nutrition in Austria
Acronym: Sukie
Status: Completed | Type: Observational
Sponsor: Karin Schindler (Other)
Responsible Party: Sponsor-Investigator, Karin Schindler, PD Dr. Karin Schindler, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: SukieAUT2019
Record Dates: First submitted 2019-10-04; First posted 2019-10-24 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Breast Feeding
Keywords: breastfeeding prevalence; infant nutrition; complimentary feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will give an update on the breastfeeding prevalence and infant nutrition in Austria.

Key aspects for this study are:

1. the current breastfeeding rates
2. further insights on factors influencing breastfeeding such as the information mothers have about breastfeeding, their attitude, support they received for breastfeeding problems as well as sociodemographic factors and
3. complimentary feeding. All postpartum women in Austria were eligible for participation. It consists of representative and prospective data recordings of breastfeeding and infant nutrition for the participating mother-child pairs via online questionnaires at four times of measurement over a period of one year.

The results of the present study will give us an update about the development of breastfeeding rates in Austria and a better understanding of entry points for interventions on child nutrition and child health.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who gave birth during the recruitment period
* Mothers older than 18 years

Exclusion Criteria:

* Teenage-mothers
* Mothers of newborns in intensive care

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Mothers who have given birth within a defined period and are aged 18 years or above.
Sampling Method: Probability Sample
Enrollment: 1666 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
Prevalence of breastfeeding after birth | Online questionnaire at 14 days postpartum (time of measurement 1)
  Proportion of mothers initiating breastfeeding: assessing the breastfeeding prevalence after birth (% of participating mothers).
Prevalence of breastfeeding | Online questionnaire at 14 days postpartum (time of measurement 1)
  Assessing the breastfeeding prevalence at 14 days postpartum (% of participating mothers)
Prevalence of breastfeeding | Online questionnaire at 4 months postpartum (time of measurement 2)
  Assessing the breastfeeding prevalence at 4 months postpartum (% of participating mothers)
Prevalence of breastfeeding | Online questionnaire at 6 months postpartum (time of measurement 3)
  Assessing the breastfeeding prevalence at 6 months postpartum (% of participating mothers)
Prevalence of breastfeeding | Online questionnaire at 12 months postpartum (time of measurement 4)
  Assessing the breastfeeding prevalence at 12 months postpartum (% of participating mothers)

SECONDARY OUTCOMES:
Duration of exclusively, predominantly or partially breastfeeding: questionnaire | Online questionnaire at 4 times of measurement within the first year of life
  The average duration of infants being breastfed exclusively, predominantly or partially at time of measurement 1 in days; at time of measurement 2-4 in months; according to the WHO indicators: proportion of infants under 6 months who are fed exclusively with breast milk, proportion of infants under 6 months who are fed predominantly with breast milk; additionally: proportion of infants under 6 months who are fed partially with breast milk
Assessment of infant feeding if breastfeeding is not performed: questionnaire | Online questionnaire at 4 times of measurement within the first year of life
  Proportion of infants receiving formula
Infant nutrition, assessment of complimentary feeding: questionnaire | Online questionnaire at 4 times of measurement within the first year of life
  Age of infant at initiation of complimentary feeding - in months; according to the WHO indicators: proportion of infants who received complementary food, proportion of infants who received 4 or more food groups
Influence of factors on breastfeeding prevalence: questionnaire | Online questionnaire at 2 times of measurement (time of measurement 1 (14 days after delivery) and 4 (12 months after delivery))
  Breastfeeding prevalence statistically dependent on socioeconomic factors and lifestyle and other general conditions - % of participating mothers
Influence of factors on breastfeeding duration: questionnaire | Online questionnaire at 2 times of measurement (time of measurement 1 (14 days after delivery) and 4 (12 months after delivery))
  Breastfeeding duration statistically dependent on socioeconomic factors, lifestyle and other general conditions: Average duration of infants being fed at time of measurement 1: in days; at time of measurement 4: in months
Structure in the maternity wards: questionnaire | One online questionnaire at study start within the recruitment period (February/March 2019)
  Proportion of participating maternity wards with BFHI certificate, offering rooming-in, providing information on breastfeeding and breastfeeding support

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna General Hospital, Vienna, Austria